CLINICAL TRIAL: NCT03805412
Title: A Pilot Study on the Use of Real-Time Continuous Glucose Monitoring (RT-CGM) as an Educational Tool for Patients With Prediabetes and Diabetes
Brief Title: Continuous Glucose Monitoring in Diabetes and Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicole Ehrhardt, MD (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Nicole Ehrhardt, MD, Endocrinologist, Principal Investigator, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 180609
Record Dates: First submitted 2018-12-19; First posted 2019-01-15 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2; PreDiabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- DEXCOM G6 RT-CGM (Active Comparator): These participants will wear blinded continuous glucose monitoring for 10 days at baseline and 14 weeks. They will also complete real-time continuous glucose monitoring (RT-CGM) for 10 days at 2 weeks and 6 weeks. They will receive Nutrition and exercise counseling at week 2 and 6. They will also receive additional training on continuous glucose monitoring.
  Interventions: Device: DEXCOM G6 RT-CGM
- Blinded CGM (No Intervention): These participants will have blinded continuous glucose monitoring(CGM) at the baseline and last 14 weeks. They will not wear continuous glucose monitoring at the interim appointments. They will receive 2 session of nutrition and exercise counseling at week 2 and 6.

INTERVENTIONS:
Device: DEXCOM G6 RT-CGM — CGM is a way to measure glucose levels in real-time. A tiny electrode called a glucose sensor is inserted under the skin to measure glucose levels in tissue fluid. A small plastic piece of tube remains inserted in the skin. It is connected to a transmitter that sits on top of the skin. It is approved for use on the abdomen for 10 days. It either records the sugars downloaded in the clinic (blinded part of the study) or it sends the information via wireless radio frequency to a monitoring/ display device or to a cellular phone so participants can see data. DEXCOM G6 is FDA approved for use in patients with diabetes and will be used in accordance with instructions as approved for diabetes.
  Arms: DEXCOM G6 RT-CGM

SUMMARY:
Evaluate the use of brief serial real time continuous monitoring (RT-CGM) as a behavior modification tool in obese patients with prediabetes and diabetes. After receiving RT-CGM, nutrition and exercise education, participants will be able to monitor their blood sugar in real time for 2 sessions . Education on how to interpret CGM in the setting of food choices and exercise coupled with nutrition and exercise information should lead to improved weight and other nutritional and exercise changes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55
2. Prediabetes (A1c 6.0-6.4) or Diabetes (A1c 7.0-10)
3. BMI ≥ 30 kg/m2
4. Willing to wear pedometer during study period
5. Able to walk 2 city blocks at baseline without assistance (self-reported)
6. Reading level at least 6th grade in English
7. Expected to remain in local community for at least 4 months
8. Either is not treated with or has been on a stable treatment regimen of any of the following medications for a minimum of 3 months prior to Visit 1 (Screening/Enrollment):

   1. Sulfonylureas
   2. Biguanidine
   3. Thyroid replacement therapy
   4. Glp-1 agonists
   5. Sodium-glucose co-transporters
   6. Basal insulin
   7. Thiazolidinediones
   8. Hormone replacement therapy (female subjects) estrogen/progesterone products
   9. Oral contraceptives/birth control (female subjects)
   10. Antidepressant agents (SSRIs, Paxil, Prozac, Celexa, Zoloft, etc.)
9. Is able to read, understand, and sign the Informed Consent Form (ICF) and if applicable, an Authorization to Use and Disclose Protected Health Information form (consistent with Health Insurance Portability and Accountability Act of 1996 [HIPAA] legislation), communicate with the investigator, and understand and comply with protocol requirements.

Exclusion Criteria:

1. Women who are pregnant, lactating, planning to become pregnant
2. Subjects who are taking amphetamines, anabolic, or weight-reducing agents
3. Contraindications to moderate exercise
4. Pre-prandial insulin
5. On any antipsychotic medication or history of schizophrenia or bipolar disorder
6. Daily use of any form of steroid medication (oral, inhaled, injected) within the last 3 months
7. Active wounds or recent surgery within 3 months
8. Inflammatory disease, or chronic and current use of anti-inflammatory drugs or narcotics
9. Active cardiovascular diseases within 12 months of Visit 1, such as myocardial infarction, clinically significant arrhythmia, unstable angina, coronary artery bypass surgery, or angioplasty; or are expected to require coronary artery bypass surgery or angioplasty during the course of the study
10. Presence or history of severe congestive heart failure (New York Heart Association Class IV [CCNYHA 1994])
11. Has evidence of current abuse of drugs or alcohol or a history of abuse that, in the investigator's opinion, would cause the individual to be noncompliant
12. Enrolled in another weight loss program
13. Already receiving continuous glucose monitoring (CGM)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Ehrhardt, MD, Principal Investigator — George Washington University
Locations (1):
- GWU Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: note study was closed early given covid so enrollement was 23 not 45 as in orginal protocol
Period: Overall Study
Arm/Group | DEXCOM G6 RT-CGM | Blinded CGM
Started | 15 | 8
Completed | 15 | 7
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DEXCOM G6 RT-CGM | Blinded CGM | Total
Number analyzed (Participants) | 15 | 8 | 23
Age, Customized [Number; unit: years]
  Participants were between the ages of 18 and 55 years old | 15 | 8 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 4 | 16
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in BMI From Baseline to 14 Weeks
Description: weight and height will be combined to report % change BMI in kg/m^2 at 14 weeks
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: % change over 14 weeks
Arm/Group | DEXCOM G6 RT-CGM | Blinded CGM
Number analyzed (Participants) | 15 | 7
% change over 14 weeks | -0.3 (0.5) | -0.2 (0.9)

2. Primary Outcome: Percent Body Fat Change at 14 Weeks
Description: Percent by Tanita scale
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: % change over 14 weeks
Arm/Group | DEXCOM G6 RT-CGM | Blinded CGM
Number analyzed (Participants) | 15 | 7
% change over 14 weeks | 1.7 (3.5) | -1.6 (3.2)

3. Secondary Outcome: Questionnaire: Experiences With Glucose Monitoring (CGM) Diabetes
Description: Experiences of CGM @Joslin 2009 scale of (5) strongly agree or (1) strongly disagree about statements/questions that measured the amount of satisfaction that was derived from continuous glucose monitoring. The larger the score the more satisfied participants were with CGM. 100 being the max score and 20 being the min score
Time Frame: 14 weeks
Population: All participants in the CGM Intervention group. Blinded group did not complete this survey
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CGM Intervention: CGM intervention group
Arm/Group | CGM Intervention
Number analyzed (Participants) | 15
score on a scale | 75.8 (9.3)

4. Secondary Outcome: Mean Glucose Change at 14 Weeks
Description: average glucose during 10 days of wearing continuous glucose monitoring (CGM) at baseline and 14 weeks
Time Frame: 14 weeks
Population: CGM average glucose(mg/dL)
Measure: Mean (Standard Deviation); unit: % change over 14 weeks
Arm/Group | DEXCOM G6 RT-CGM | Blinded CGM
Number analyzed (Participants) | 15 | 7
% change over 14 weeks | -0.3 (28.9) | 23.0 (61.9)

5. Secondary Outcome: Food Frequency Change in Score at 14 Weeks
Description: Starting The Conversation (STC) is an eight-item simplified food frequency instrument/questionnaire a max score of 16 indicates poor food choices and a minimum score of 0 indicates good food choices. Results reported is change from baseline score with a negative score being a marker of improvement in food choices and a positive score being worsening of food choices
Time Frame: 14 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | DEXCOM G6 RT-CGM | Blinded CGM
Number analyzed (Participants) | 15 | 7
score on a scale | -2.0 [-2.8 to 0.2] | 0 [-1.2 to 1.6]

6. Secondary Outcome: Change in Minutes Walked Per Week at 14 Weeks
Description: The International Physical Activity Questionnaire(short) is as validated questionnaire which asks the time in minutes or hours in last week you do vigorous exercise, moderate intensity exercise, walking and sitting
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: minutes walked per week
Arm/Group | DEXCOM G6 RT-CGM | Blinded CGM
Number analyzed (Participants) | 15 | 7
minutes walked per week | 438.8 (535.4) | 232.0 (343.6)

7. Secondary Outcome: MAGE Mean Amplitude of Glycemic Excursion
Description: this is calculation of variance of glucose for CGM
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: mg/100ml
Arm/Group | DEXCOM G6 RT-CGM | Blinded CGM
Number analyzed (Participants) | 15 | 7
mg/100ml | 95.1 (32.3) | 90.1 (85.9)
Statistical Analysis 1: Comparison: DEXCOM G6 RT-CGM vs Blinded CGM; Test type: Superiority; p = 0.694, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 14 weeks
Arm/Group | DEXCOM G6 RT-CGM | Blinded CGM
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/8
Other Adverse Events (participants affected / at risk) | 0/15 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT03805412/Prot_001.pdf
  • Statistical Analysis Plan (2018-11-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT03805412/SAP_003.pdf